CLINICAL TRIAL: NCT01581203
Title: A Phase 3 Study With Asunaprevir and Daclatasvir (DUAL) for Null or Partial Responders to Peginterferon Alfa and Ribavirin (P/R), Intolerant or Ineligible to P/R Subjects and Treatment-Naive Subjects With Chronic Hepatitis C Genotype 1b Infection
Brief Title: Phase III Hallmark DUAL: ASV+DCV (Nulls/Partials, Intolerants/Ineligibles. Naives)
Acronym: Hallmark DUAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AI447-028; 2011-005446-35 (EudraCT Number)
Record Dates: First submitted 2012-04-18; First posted 2012-04-20 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — asunaprevir; daclatasvir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1: Null or Partial Responder to P/R (ASV + DCV) (Experimental): Asunaprevir 100 mg Capsules by mouth, Twice daily for 24 Weeks
  Daclatasvir 60 mg Tablet by mouth, Once daily for 24 Weeks
  Interventions: Drug: Asunaprevir (ASV); Drug: Daclatasvir (DCV)
- Arm 2: Intolerant to or Ineligible for P/R (ASV + DCV) (Experimental): Asunaprevir 100 mg Capsules by mouth, Twice daily for 24 Weeks
  Daclatasvir 60 mg Tablet by mouth, Once daily for 24 Weeks
  Interventions: Drug: Asunaprevir (ASV); Drug: Daclatasvir (DCV)
- Arm 3: Treatment naive (ASV + DCV) (Experimental): [Subjects will receive ASV + DCV for 24 weeks] followed by ASV + DCV for 24 weeks in protocol AI444026]
  Subjects meeting prespecified rescue criteria in the treatment naive cohort may have therapeutic rescue instituted with QUAD regimen (QUAD= ASV + DCV + P/R)
  Asunaprevir 100 mg Capsules by mouth, Twice daily for 24 or 48 Weeks
  Daclatasvir 60 mg Tablet by mouth, Once daily for 24 or 48 Weeks
  Pegylated-interferon alfa 2a (PegIFN) 180 mcg/0.5 mL injection subcutaneously (SC), once weekly for 24 or 48 weeks
  Ribavirin 1000 mg/1200 mg (total daily dose) tablet by mouth for 24 or 48 weeks
  Interventions: Drug: Asunaprevir (ASV); Drug: Daclatasvir (DCV); Drug: Pegylated-interferon alfa 2a (PegIFN); Drug: Ribavirin (RBV)
- Arm 4: Null or Partial Responder to P/R (ASV + DCV) 24/48 week (Experimental): Subjects meeting prespecified rescue criteria in the null or partial responder cohort or active arm of the treatment naive cohort may have therapeutic rescue instituted with QUAD regimen (QUAD= ASV + DCV + P/R)
  Asunaprevir 100 mg Capsules by mouth, Twice daily for 24 or 48 Weeks
  Daclatasvir 60 mg Tablet by mouth, Once daily for 24 or 48 Weeks
  Pegylated-interferon alfa 2a (PegIFN) 180 mcg/0.5 mL injection subcutaneously (SC), once weekly for 24 or 48 weeks
  Ribavirin 1000 mg / 1200 mg (total daily dose) Tablet by mouth, for 24 or 48 weeks
  Interventions: Drug: Asunaprevir (ASV); Drug: Daclatasvir (DCV); Drug: Pegylated-interferon alfa 2a (PegIFN); Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: Asunaprevir (ASV)
  Other Names: BMS-650032
Drug: Daclatasvir (DCV)
  Other Names: BMS-790052
Drug: Pegylated-interferon alfa 2a (PegIFN)
  Other Names: Pegasys
  Arms: Arm 3: Treatment naive (ASV + DCV); Arm 4: Null or Partial Responder to P/R (ASV + DCV) 24/48 week
Drug: Ribavirin (RBV)
  Other Names: Copegus
  Arms: Arm 3: Treatment naive (ASV + DCV); Arm 4: Null or Partial Responder to P/R (ASV + DCV) 24/48 week

SUMMARY:
The purpose of this study is to estimate efficacy, as determined by the proportion of subjects with Sustained virologic response at post-treatment Week 12 (SVR12), defined as Hepatitis C virus (HCV) Ribonucleic acid (RNA) < Limit of quantitation (LOQ) at post-treatment Week 12, for subjects who are prior null or partial responders to P/R or who are treatment-naive.

DETAILED DESCRIPTION:
Allocation: Treatment naive cohort: Randomized Controlled Trial, Null/partial responder and intolerant/ineligible cohorts: N/A (Single arm study)

Masking: Treatment naive cohort: Double Blind, Null/partial responder and intolerant/ineligible cohorts: Open

Intervention Model: Treatment naive cohort: Parallel, Null/partial responder and intolerant/ineligible cohorts: Single group

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Males and females, ≥ 18 years of age
* HCV Genotype 1b who previously failed treatment with peginterferon alfa and ribavirin, classified as previous null or partial responders based on previous therapy, OR intolerant or ineligible to P/R due to neutropenia, anemia, depression or thrombocytopenia with fibrosis/cirrhosis, OR treatment naive
* HCV RNA ≥ 10,000 IU/mL
* Seronegative for Human immunodeficiency virus (HIV) and Hepatitis B surface antigen (HBsAg)
* Subjects with compensated cirrhosis are permitted (compensated cirrhotics are capped at approximately 25% of treated population)

Exclusion Criteria:

* Prior treatment of HCV with HCV direct acting antiviral (DAA)
* Evidence of a medical condition contributing to chronic liver disease other than HCV
* Evidence of decompensated liver disease including, but not limited to, a history or presence of ascites, bleeding varices, or hepatic encephalopathy
* Diagnosed or suspected hepatocellular carcinoma or other malignancies
* Uncontrolled diabetes or hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 748 (Actual)
Dates: Start 2012-05; Primary Completion 2013-10 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Proportion of treated subjects with SVR12, defined as HCV RNA < LOQ at post treatment Week 12, for subjects who are prior null or partial responders to P/R or are treatment-naive | At 12 weeks post-treatment

SECONDARY OUTCOMES:
Proportion of treated subjects with SVR12, defined as HCV RNA < LOQ at post-treatment Week 12, for subjects who are intolerant or ineligible to P/R | Post-treatment Week 12
On treatment safety, as measured by frequency of Serious Adverse Events (SAEs) and discontinuations due to Adverse Events (AEs) | End of Treatment (up to 48 weeks) plus 7 days
Differences in rates of selected grade 3-4 laboratory abnormalities during the first 12 weeks between treatments (ASV + DCV vs PBO) for naive subjects | Up to first 12 weeks
Proportion of genotype 1b subjects with SVR12 (HCV RNA < LOQ at post treatment Week 12) by the rs12979860 single nucleotide polymorphisms (SNP) in the IL28B gene for each cohort | Post-treatment Week 12
Proportion of genotype 1b subjects with HCV RNA undetectable | At weeks 1, 2, 4, 6, 8 and 12; at both Weeks 4 and 12 [eRVR]; EOT (up to 24 weeks), post-treatment Week 12, or post-treatment Week 24 for each cohort
  eRVR = Extended rapid virologic response, EOT = End of treatment
Proportion of genotypes 1b subjects with HCV RNA < LOQ | At weeks 1, 2, 4, 6, 8 and 12; at both Weeks 4 and 12 [VR(4&12)]; EOT (up to 24 weeks), post-treatment Week 24 (SVR24) for each cohort
Proportion of subjects with anemia | At 12 weeks post-treatment
Proportion of subjects with rash | At 12 weeks post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (100):
- United States (18):
  - The Health Care Authority For Baptist Health, Montgomery, Alabama
  - Scripps Clinic, La Jolla, California
  - Scpmg/ Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - University Of Colorado Denver And Hospital, Aurora, Colorado
  - Uf Hepatology Research At Ctrb, Gainesville, Florida
  - Johns Hopkins Medical Institutions, Lutherville, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Washington University School Of Medicine, St Louis, Missouri
  - North Shore-Long Island Jewish Health System, Manhasset, New York
  - Weill Cornell Medical College, New York, New York
  - University Of North Carolina At Chapel Hill School Of Med, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Baylor College Of Medicine, Houston, Texas
  - Vamc, Houston, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Dean Clinic, Madison, Wisconsin
- Argentina (3):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Ciudad de Buenos Aires, Buenos Aires
  - Local Institution, Prov de Santa Fe, Santa Fe Province
- Australia (12):
  - Local Institution, Darlinghurst, New South Wales
  - Local Institution, Kogarah, New South Wales
  - Local Institution, Randwick, New South Wales
  - Local Institution, Fitzroy, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Bedford Park, Sa, South Australia
  - Local Institution, Clayton, Victoria
  - Local Institution, Heidelberg, Victoria
  - Local Institution, Melbourne, Victoria
  - Local Institution, Fremantle, Western Australia
  - Local Institution, Nedlands, Western Australia
  - Local Institution, Perth, Western Australia
- Austria (4):
  - Local Institution, Graz
  - Local Institution, Linz
  - Local Institution, Salzburg
  - Local Institution, Vienna
- Canada (8):
  - Gastrointestinal Research Institute (G.I.R.I.), Vancouver, British Columbia
  - Percuro Clinical Research Ltd, Victoria, British Columbia
  - Toronto General Hospital-University Health Network, Toronto, Ontario
  - Toronto Liver Centre, Toronto, Ontario
  - Toronto Digestive Disease Associates, Inc., Vaughan, Ontario
  - Clinique Medicale Lactuel, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Alpha-Recherche Clinique, Québec, Quebec
- France (7):
  - Local Institution, Clichy
  - Local Institution, Créteil
  - Local Institution, Lyon
  - Local Institution, Marseille
  - Local Institution, Paris
  - Local Institution, Toulouse
  - Local Institution, Vandœuvre-lès-Nancy
- Germany (7):
  - Local Institution, Berlin
  - Local Institution, Bonn
  - Local Institution, Essen
  - Local Institution, Frankfurt
  - Local Institution, Hamburg
  - Local Institution, Hanover
  - Local Institution, München
- Local Institution, Dublin, Dublin, Ireland
- Israel (5):
  - Local Institution, Haifa
  - Local Institution, Jerusalem
  - Local Institution, Tel Aviv
  - Local Institution, Tel Litwinsky
  - Local Institution, Zafed
- Italy (4):
  - Local Institution, Messina
  - Local Institution, Milan
  - Local Institution, Roma
  - Local Institution, Torino
- Netherlands (3):
  - Local Institution, Amsterdam
  - Local Institution, Leiden
  - Local Institution, Rotterdam
- New Zealand (3):
  - Local Institution, Auckland
  - Local Institution, Hamilton
  - Local Institution, Wellington
- Poland (2):
  - Local Institution, Bialystok
  - Local Institution, Wroclaw
- Russia (7):
  - Local Institution, Chelyabinsk
  - Local Institution, Krasnoyarsk
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
  - Local Institution, Samara
  - Local Institution, Smolensk
  - Local Institution, Tyumen
- South Korea (6):
  - Local Institution, Busan
  - Local Institution, Daegu
  - Local Institution, Gyeonggi-do
  - Local Institution, Gyeongsangnam-do
  - Local Institution, Incheon
  - Local Institution, Seoul
- Spain (4):
  - Local Institution, Alicante
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Valencia
- Taiwan (3):
  - Local Institution, Taichung
  - Local Institution, Tainan
  - Local Institution, Taipei
- United Kingdom (3):
  - Local Institution, London, Greater London
  - Local Institution, Manchester, Greater Manchester
  - Local Institution, Glasgow, Lanarkshire

REFERENCES:
- [Derived] Kao JH, Lee YJ, Heo J, Ahn SH, Lim YS, Peng CY, Chang TT, Torbeyns A, Hughes E, Bhore R, Noviello S. All-oral daclatasvir plus asunaprevir for chronic hepatitis C virus (HCV) genotype 1b infection: a sub-analysis in Asian patients from the HALLMARK DUAL study. Liver Int. 2016 Oct;36(10):1433-41. doi: 10.1111/liv.13128. Epub 2016 Apr 28. PMID 27009831
- [Derived] Kao JH, Jensen DM, Manns MP, Jacobson I, Kumada H, Toyota J, Heo J, Yoffe B, Sievert W, Bessone F, Peng CY, Roberts SK, Lee YJ, Bhore R, Mendez P, Hughes E, Noviello S. Daclatasvir plus asunaprevir for HCV genotype 1b infection in patients with or without compensated cirrhosis: a pooled analysis. Liver Int. 2016 Jul;36(7):954-62. doi: 10.1111/liv.13049. Epub 2016 Jan 24. PMID 26683763
- [Derived] Manns M, Pol S, Jacobson IM, Marcellin P, Gordon SC, Peng CY, Chang TT, Everson GT, Heo J, Gerken G, Yoffe B, Towner WJ, Bourliere M, Metivier S, Chu CJ, Sievert W, Bronowicki JP, Thabut D, Lee YJ, Kao JH, McPhee F, Kopit J, Mendez P, Linaberry M, Hughes E, Noviello S; HALLMARK-DUAL Study Team. All-oral daclatasvir plus asunaprevir for hepatitis C virus genotype 1b: a multinational, phase 3, multicohort study. Lancet. 2014 Nov 1;384(9954):1597-605. doi: 10.1016/S0140-6736(14)61059-X. Epub 2014 Jul 28. PMID 25078304
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx